CLINICAL TRIAL: NCT06724380
Title: Detection of Health Risk Situations in the Anesthesia Consultation.
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-64
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: unknown health risk situation — a unknown health risk situation detected at anestesiology consult

SUMMARY:
This study aims to estimate the proportion of patients seen in the anesthesiology consultation for planned surgery in whom a previously unknown health risk situation is detected (e.g., obesity, anemia, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 50 years.

  * Indication for elective surgery.
  * In-person preoperative evaluation in the scheduled Anesthesiology consultation.

Exclusion Criteria:

* Indication for non-deferrable urgent surgery.
* Pregnant women.
* Pre-surgical visit outside the anesthesia consultation.
* Incomplete preoperative evaluation, as indicated in the final section (preoperative judgment) of the anesthesia visit report.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients evaluated in person at the preoperative anesthesia consultation for a scheduled surgery indication.
Sampling Method: Non-Probability Sample
Enrollment: 218 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
unknown health risk situation | 1 year
  proportion of patients with a unknown health risk situation

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari Alt Penedés-Garraf, Vilafranca Del Penedés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.